CLINICAL TRIAL: NCT05869266
Title: A Prospective, Crossover Randomized Controlled Trial to Compare Subjective Outcome of a Self-fitting Process Using Tuned App to a Licensed Professional Fitting
Brief Title: Tuned App Self-Fitting vs. Professional Fitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuned Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TU1-PLN-111
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hearing Loss
Keywords: self fitting
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Prospective, randomized crossover clinical study comparing two methods of fitting subjects with mild to moderate sensorineural hearing loss with hearing aids. Subjects will receive hearing aids and be assigned to professional-fitting arm or self-fitting arm, use the hearing aids for two weeks then switch to the other arm and use the hearing aids for another two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Professional-fitting (Active Comparator): Subject receives hearing aids and a licensed professional performs the hearing aid fitting using professional programing tools, and the thresholds that were obtained from the traditional audiometry.
  Subject uses the professionally fitted hearing aids for two weeks then completes COSI and the IOI-HA questionnaires.
  Interventions: Device: professional fitting vs. self fitting
- Self-fitting (Active Comparator): Subject receives hearing aids, downloads the Tuned self fitting App and performs self-fitting of the hearing aids including a self-hearing test.
  Subject uses the self fitted hearing aids for two weeks then completes COSI and the IOI-HA questionnaires.
  Interventions: Device: professional fitting vs. self fitting

INTERVENTIONS:
Device: professional fitting vs. self fitting — Licensed professional fits the hearing aid fitting using professional programing tools and thresholds obtained from the traditional audiometry vs. subject performs self-fitting of the hearing aids using the Tuned App.
  Other Names: Tuned App

SUMMARY:
The aim of the study is to compare the perceived outcome of the self-fitting performed by the participants using the Tuned mobile application with the traditional professional fitting as performed by a licensed professional audiologist in subjects with mild to moderate sensorineural hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, 18 years and older.
* Mild to moderate sensorineural hearing loss.
* Own and able to use a smart phone (Android or iOS).
* Able to read and understand Hebrew.

Exclusion Criteria:

* Conductive mixed hearing loss.
* Unilateral hearing loss.
* Any external or inner ear malformations.
* Symptoms of ear disease or excessive cerumen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Comparison of self fitting and professional fitting by COSI scores | 4 weeks
  To compare the professional fitting and the self fitting using the Tuned App, the scores of Client Oriented Scale of Improvement (COSI) questionnaire will be used.

SECONDARY OUTCOMES:
Comparison of self fitting and professional fitting by IOI-HA scores | 4 weeks
  To compare the subjects' self-reported outcomes between professional fitting and self fitting using the Tuned App, the scores of the International Outcome Inventory for Hearing Aids (IOI-HA) questionnaires will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Kriksunov, Principal Investigator — Ozen-Kashevet Hearing Clinic
Locations (1):
- Ozen-Kashevet Hearing Clinic, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided